CLINICAL TRIAL: NCT01958190
Title: A Multicenter Randomized in Primary Livertransplantation Comparing Longterm Renal Function in Recipients Treated With Tacrolimus Alone and Recipients Treated With a Combination Tacrolimus and Sirolimus
Brief Title: Study Comparing in Livertransplantation Recipients With Tacrolimus Alone Versus Tacrolimus&Sirolimus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOL-III-1
Record Dates: First submitted 2013-08-27; First posted 2013-10-09 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Liver Disease
Keywords: Liver transplantation long term renal function; tacrolimus sirolimus
MeSH Terms: conditions — Liver Diseases | interventions — Tacrolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus (Active Comparator): Patient received standard-dose of Tracrolimus Advagraf (5-10 ng/ml) and 7.5 mg prednison; lower or discontinue steroids after day 180 at the discretion of the treating physician
  Interventions: Drug: Tacrolimus
- combination Tacrolimus and Sirolimus (Experimental): Patients receive combination of low-dose extended release Tacrolimus and low-dose Sirolimus
  Interventions: Drug: Tacrolimus and Sirolimus

INTERVENTIONS:
Drug: Tacrolimus and Sirolimus — Arm 1 once daily combination therapy of normal dosed extended-release tacrolimus and prednisone for 3 months and monotherapy once daily extended-release tacrolimus thereafter up to 3 years after liver transplantation.
  Arm 2 once daily combination therapy of low doses sirolimus and extended-release tacrolimus and prednisone for 3 months and combination therapy of low dose sirolimus and extended-release tacrolimus thereafter for up to 3 years after liver transplantation Continue Advagraf (5-10 ng/ml) and 7.5 mg prednison; lower or discontinue steroids after day 180 at the discretion of the treating physician Conversion to sirolimus (3-5 ng/ml) and decrease Advagraf (3-5 ng/ml); 7.5 mg prednisone and lower or discontinue steroids after day 180 at the discretion of the treating physician
  Other Names: Advagraf [Astellas Pharma bv); Rapamune
  Arms: combination Tacrolimus and Sirolimus
Drug: Tacrolimus — Patient received standard-dose of Tracrolimus Advagraf (5-10 ng/ml) and 7.5 mg prednison; lower or discontinue steroids after day 180 at the discretion of the treating physician
  Other Names: Advagraf
  Arms: Tacrolimus

SUMMARY:
In this study we compare long term renal function in liver transplantation recipients treated with standard dose extended-release tacrolimus alone and recipients treated with a combination of low dose extended-release tacrolimus and low dose sirolimus. The hypothesis is that the patients treated with the combination have better long term renal function than the patients treated with standard dose tacrolimus alone.

DETAILED DESCRIPTION:
To evaluate the effectiveness and safety of concentration controlled combination of once daily dosed low-dose sirolimus (trough levels: 3-5 ng/ml) and extended-release tacrolimus (trough levels:3-5 ng/ml), in order to provide superior renal function while maintaining comparable rates of patient and graft survival, compared to concentration controlled once - daily extended release tacrolimus (trough levels: 5-10 ng/ml) at 12, 24 and 36 months post-transplant. Moreover, to compare the incidence of de novo malignancy, the quality of life, fatigue and side effects between both treatment arms.

2.1 Primary objectives: To evaluate the effectiveness and safety of concentration controlled combination of low-dose sirolimus (trough levels: 3-5 ng/ml) and extended-release tacrolimus (trough levels: 3-5 ng/ml), in order to provide superior renal function while maintaining comparable rates of patient and graft survival, compared to concentration controlled once - daily extended release tacrolimus (trough levels:-10 ng/ml) control at 12, 24 and 36 months post-transplant.

2.2. Secondary objectives:

* To compare the incidence of de novo and recurrence of cancer between study arm and control arm at 36 months.
* To compare the incidence and severity of biopsy proven acute rejection between study arm and control arm at 12, 24 and 36 months.
* To evaluate renal function at 12, 24 and 36 months (calculated GFR).
* To evaluate the development of new onset diabetes mellitus at 12, 24 and 36 months post transplant
* To evaluate the prevalence of CNI side effects at 12, 24 and 36 months
* To evaluate quality of life (Eq5D) and fatigue severity score at 12, 24 and 36 months
* To evaluate the percentage of patients on combination tacrolimus and sirolimus and converted back to tacrolimus mono-therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary liver transplantation or retransplantation within 14 days after first transplantation
* Use of Advagraf at least 2 weeks prior to randomization
* Patent hepatic artery
* Closed abdominal wound
* Stable graft function
* Positive informed consent at time of randomization
* Age 18-70 years

Exclusion Criteria:

* Treatment with investigational drugs within 3 months before start of therapy
* Multi organ transplantation
* cGFR < 30 ml/min
* Proteinuria > 800 mg/24 h
* Hyperlipidemia refractory to optimal medical management (Cholesterol > 9 mmol/l and/or triglycerides > 8.5 mmol/l). Patients with controlled hyperlipidemia are acceptable at the time of randomization.
* Known hypersensitivity to sirolimus or its derivatives
* Thrombocytes < 50 x 109 /L
* Leukocytes < 2.5 x 109 /L
* Haemoglobin < 6 mmol/L
* Biopsy proven rejection 2 weeks prior to randomization
* HIV positivity
* Signs of recurrent or de novo cancer
* Patients with non-HCC malignancies within the past 5 years (excluding successfully treated squamous cell carcinoma and basal cell carcinoma of the skin)
* Evidence of significant local or systemic infection
* Pregnancy or breast feeding
* Women of child-bearing potential not willing to take oral contraception
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-02-07 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Renal function | 3 years
  Percentage of patients with cGFR < 60ml/min

SECONDARY OUTCOMES:
Malignancies | 3 years
  number of de novo malignancies
Diabetes Mellitus | 3 years
  Incidence of De novo diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Herold J Metselaar, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - UMCG, Groningen
  - LUMC, Leiden
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided